CLINICAL TRIAL: NCT07357103
Title: Positioning Second-line Therapies for Pneumocystis Jirovecii Pneumonia (PCP Alternatives) [A Branch of the Initial Treatment Domain of the SPIRIT-PCP Platform]
Brief Title: Positioning Second-line Therapies for Pneumocystis Jirovecii Pneumonia (PCP Alternatives)
Acronym: SPIRIT-ALT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Associate professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026-12268; 527077 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-12-27; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Pneumocystis; Pneumocystis Infection; Pneumocystis Carinii Infection; Pneumocystis Carinii; Infection, Resulting From HIV Disease; Pneumocystis Jirovecii Pneumonia; Pneumocystis Jirovecii Infection; Pneumocystosis Associated With AIDS; Pneumocystosis; Pneumonia (Etiology)
Keywords: PCP; Pneumocystis jirovecii pneumonia; PCP Alternatives; Clindamycin; Pentamidine; Primaquine; Atovaquone; HIV; Non-HIV; Immunocompromised host; Randomized Control Trial
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumocystis Infections; Infections; Pneumonia | interventions — Clindamycin; Primaquine; Pentamidine; Atovaquone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Severe PCP-Clindamycin+primaquine (Experimental): Participants with severe PCP will be randomized to receive clindamycin in combination with primaquine as second-line therapy due to intolerance of or contraindications to trimethoprim-sulfamethoxazole.
  Interventions: Drug: Clindamycin + primaquine
- Severe PCP-Intravenous Pentamidine (Experimental): Participants with severe PCP will be randomized to receive intravenous pentamidine as second-line therapy due to intolerance of or contraindications to trimethoprim-sulfamethoxazole.
  Interventions: Drug: Pentamidine
- Mild to Moderate PCP- Clindamycin+primaquine (Experimental): Participants with mild to moderate PCP will be randomized to receive clindamycin in combination with primaquine as second-line therapy due to intolerance of or contraindications to trimethoprim-sulfamethoxazole.
  Interventions: Drug: Clindamycin + primaquine
- Mild to moderate PCP- Atovaquone (Experimental): Participants with mild to moderate PCP will be randomized to receive atovaquone as second-line therapy due to intolerance of or contraindications to trimethoprim-sulfamethoxazole.
  Interventions: Drug: Atovaquone

INTERVENTIONS:
Drug: Clindamycin + primaquine — Participants randomized to this intervention will receive clindamycin in combination with primaquine as second-line therapy for the treatment of PCP.
  This regimen may be used for participants with Severe PCP or mild to moderate PCP in acccordance with protocol-defined disease severity and standard clinical practice.
  Arms: Mild to Moderate PCP- Clindamycin+primaquine; Severe PCP-Clindamycin+primaquine
Drug: Pentamidine — Participants randomized to this intervention will receive pentamidine, administered intravenously, as second-line therapy for the treatment of PCP in patients with severe disease who are unable to tolerate or have contraindications to trimethoprim-sulfamethoxazole (TMP/SMX)
  Arms: Severe PCP-Intravenous Pentamidine
Drug: Atovaquone — Participants randomized to. this intervention will receive atovaquone, administered orally, as second-line therapy for the treatment of PCP in participants with mild to moderate disease who are unable to tolerate or have contraindications to trimethoprim-sulfamethozaxole (TMP/SMX).
  Arms: Mild to moderate PCP- Atovaquone

SUMMARY:
The usual first treatment for Pneumocystis jirovecii pneumonia (PCP) is an antibiotic called trimethoprim-sulfamethoxazole (TMP-SMX). However, some patients cannot take this medication because of allergies, side effects, or lack of response.

This study asks the question:

When TMP-SMX cannot be used, which alternative treatment for PCP provides the best balance of effectiveness and safety?

DETAILED DESCRIPTION:
Pneumocystis jirovecii pneumonia (PCP) is a serious lung infection that affects people with weakened immune systems (e.g., patients with cancer, organ transplants, autoimmune diseases, or HIV). Without timely treatment, PCP can lead to respiratory failure and death.

TMP-SMX is the standard first-line treatment, but 20-30% of patients cannot receive the treatment or cannot tolerate it due to allergic reactions, kidney problems, low blood counts, drug interactions, or treatment failure. In these situations, doctors use alternative medications such as clindamycin with primaquine, pentamidine, or atovaquone.

Although these alternative treatments are widely used, there is limited modern research directly comparing them. As a result, treatment choices vary between hospitals and physicians.

The main objective of this study is to determine which alternative treatment works best for patients with PCP who cannot receive TMP-SMX. Eligible participants in the PCP alternatives therapy are enrolled and randomized centrally 1:1 in the MUHC Research Electronic Data Capture (REDCap) system. The primary outcome is a Hierarchical composite Win Ratio Outcome at day 30: death; new extracorporeal membrane oxygenation (ECMO), new invasive mechanical ventilation; severe (CTCAE grade 4) adverse drug event; and length of stay in hospital (amongst survivors). Secondary endpoints include individual components of the composite outcome, and tertiary endpoints include quality of life and longer-term outcomes through day 180.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patients (including but not limited to HIV, solid organ transplant, solid tumors, hematological transplant and malignancies, systemic diseases, chemotherapy, long term corticosteroid use, and immunosuppressive therapies, as well as primary immunodeficiencies) in an emergency department, cliinic, or hospital

  * Age ≥18 years
  * Proven or probable Pneumocystis jirovecii pneumonia
  * Inability to receive trimethoprim-sulfamethoxazole due to contraindication, intolerance, toxicity, or treatment failure
  * Immunocompromised status
  * Ability to provide informed consent (or per local regulations)

While participants may be enrolled in multiple domains of the SPIRIT-PCP Platform over time (if they are eligible and a domain is active), they may only be enrolled to single question once (e.g., they can be part PCP Alternatives and an eventual secondary prophylaxis domain; however, if they have a recurrence, they cannot be included in PCP Alternatives again).

Exclusion Criteria:

* The Platform will exclude: patients where we are unable to obtain informed consent, where patients or their proxy have declined to consent, where the treating team has declined participation, where follow up cannot be reliably obtained (e.g., lack of means of communication, patient non-resident of jurisdiction), where treatment with antibiotics is not in keeping with a patient's advanced care directives, and where death is deemed imminent (<48h) as determined by the treating team and site investigator.

Clinical:

1. Previous severe adverse reaction or hypersensitivity to clindamycin, primaquine, or atovaquone (mild-moderate PCP) or to clindamycin, primaquine, or pentamidine (severe PCP);
2. More than 7 calendar days of any therapy for PCP (no more than 4 can involve a study drug).
3. Known pregnancy or breastfeeding (pregnancy test will be offered)

   Drug specific exclusion criteria:
4. For clindamycin-primaquine:

   1. Known G6PD deficiency OR family history of G6PD deficiency without excluding by testing*
   2. Known diagnosis of porphyria
   3. Concomitant use of methotrexate or cyclophosphamide which cannot be held *G6PD deficiency is an X-linked recessive genetic disease. Female patients without a family history are very unlikely to have this disease and so therapy can start while waiting for the test in the absence of a family history. Male patients should wait for test results prior to receiving primaquine even if they do not have a family history. For those without G6PD testing at diagnosis, it is a reasonable standard of care to order testing.
5. For pentamidine:

   1. Absence of adequate intravenous access as determined by treating team and site investigator. In the event of loss of IV, up to 2 consecutive doses can be given intramuscularly if the patient is not systemically anticoagulated and does not have a coagulopathy.
   2. Hypotension defined as systolic blood pressure below 90mmHg without pharmacologic support
   3. Personal history of Torsade de Pointes or presence of a corrected QTc of greater than 490ms on ECG on date of enrollment
6. For atovaquone:

   1. Receipt of PCP Prophylaxis (≥3 doses per week) for ≥ 4 weeks with atovaquone
   2. inability to tolerate atovaquone with a meal or enteral feeding (e.g., prolonged NPO status is an exclusion as atovaquone must be taken with food for proper absorption)
   3. Concurrent use of rifampin, rifabutin, or tetracycline (that cannot be stopped)
   4. Reduced gastric absorption (patient must not have a medical condition which the treating team and/or site investigator believes will interfere with atovaquone absorption, e.g., total gastrectomy)

Administrative:

1. Trial site not participating in PCP Alternatives branch of the initial therapy domain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite outcome | Day 30
  Hierarchical composite of Win Ratio at day 30:
  * death;
  * new extracorporeal membrane oxygenation (ECMO),
  * new invasive mechanical ventilation;
  * severe (CTCAE grade 4) adverse drug event (dermatologic, nephrologic, hematologic, neurologic, and/or endocrinologic) considered at least probable (by Leape and Bates criteria);
  * new non-invasive ventilation;
  * change of therapy (i.e., dose or agent) due to presumed treatment failure or probable adverse drug reaction (by Leape and Bates criteria); and
  * length of stay in hospital (amongst survivors)

SECONDARY OUTCOMES:
Proportion of patients that die (death) | Day 30
  Mortality at day 30
Proportion of patients with a need for new extracorporeal membrane oxygenation (ECMO), | Day 30
  New initiation of extracorporeal membrane oxygenation during hospitalization following initiation of assigned PCP treatment strategy.
Proportion of patients requiring new Invasive Mechanical Ventilation | Day 30
  Initiation of invasive mechanical ventilation via endotracheal intubation during hospitalization following initiation of the assigned PCP treatment strategy.
Proportion of patients with severe (CTCAE grade 4) adverse drug event | Day 30
  Proportion of patients with occurence of severe (CTCAE grade 4) adverse drug event (dermatologic, nephrologic, hematologic, neurologic, and/or endocrinologic) considered at least probable (by Leape and Bates criteria).
Proportion of patients with need for new non-invasive ventilation; | Day 30
  initiation of non-invasive ventilation (including continuous positive airway pressure [CPAP] or bilevel positive airway pressure [BiPAP] during hospitalization following initiation of the assigned PCP treatment strategy.
Proportion of patients requiring escalation or change of PCP -directed therapy | Day 30
  Proportion of patients with escalation or change of PCP -directed therapy due to inadequate clinical response, disease progression, or treatment-limiting toxicity during the treatment or follow-up period.
Median length of stay in hospital amongst survivors | Day 30
  Length of hospital stay, measured in days from hospital admission to discharge among participants who survive to hospital discharge.

OTHER OUTCOMES:
Tertiary outcome measure of quality of life at day 30 | Day 30
  Quality of life (EQ-5D-5L) wherein a higher score indicates better quality of life.
Tertiary outcome measure of all-cause mortality | Day 180
  All-cause mortality, defined as death from any cause.
Tertiary Outcome Measure of PCP recurrence | Day 180
  Recurrence of pneumocystis pneumonia, defined as a new episode of clinically and/or microbiologically confirmed PCP after initial resolution.
Tertiary Outcome measure of quality of life at day 180 | Day 180
  Quality of life assessed using a EQ-5D-5L questionnaire. High score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emily G McDonald, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Todd C Lee, MD MPH, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Matthew P Cheng, MD FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized patient data will be shared for one year, released one year following the publication of the primary PCP Alternatives Manuscript. Data will be accessible through reasonable request to Emily McDonald at emily.mcdonald@mcgill.ca and with an inter-institutional agreement in place.
Access Criteria: Contact emily.mcdonald@mcgill.ca; scientists seeking to answer secondary questions about the data or combine the data in a systematic review or meta-analysis. They can access anonymous individual patient data. There will need to be an inter-institutional data sharing agreement in place.

REFERENCES:
- [Result] Del Corpo O, Butler-Laporte G, Sheppard DC, Cheng MP, McDonald EG, Lee TC. Diagnostic accuracy of serum (1-3)-beta-D-glucan for Pneumocystis jirovecii pneumonia: a systematic review and meta-analysis. Clin Microbiol Infect. 2020 Sep;26(9):1137-1143. doi: 10.1016/j.cmi.2020.05.024. Epub 2020 May 30. PMID 32479781
- [Result] McDonald EG, Afshar A, Assiri B, Boyles T, Hsu JM, Khuong N, Prosty C, So M, Sohani ZN, Butler-Laporte G, Lee TC. Pneumocystis jirovecii pneumonia in people living with HIV: a review. Clin Microbiol Rev. 2024 Mar 14;37(1):e0010122. doi: 10.1128/cmr.00101-22. Epub 2024 Jan 18. PMID 38235979
- [Result] McDonald EG, Butler-Laporte G, Del Corpo O, Hsu JM, Lawandi A, Senecal J, Sohani ZN, Cheng MP, Lee TC. On the Treatment of Pneumocystis jirovecii Pneumonia: Current Practice Based on Outdated Evidence. Open Forum Infect Dis. 2021 Oct 29;8(12):ofab545. doi: 10.1093/ofid/ofab545. eCollection 2021 Dec. PMID 34988242